CLINICAL TRIAL: NCT04765215
Title: Investigation of the Effectiveness of CoronaVac Vaccine in Cancer Patients With Active Chemotherapy and Comparison With Healthy People.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asoc. Prof. Erdoğan Selçuk Şeber (Other)
Responsible Party: Sponsor-Investigator, Asoc. Prof. Erdoğan Selçuk Şeber, Namik Kemal University (BAP), Namik Kemal University
Organization: Namik Kemal University (Other)
Other Study IDs: CHEMOCOVAC
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Is the Coronovac Vaccine Effective in Patients Receiving Chemotherapy
Keywords: coronovac; covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast or lung cancer patients receiving active chemotherapy and 2 doses of CoronaVac vaccine
  Interventions: Biological: CoronoVAC
- Healthy volunteers who received two doses of coronavac vaccine
  Interventions: Biological: CoronoVAC

INTERVENTIONS:
Biological: CoronoVAC — SARS-CoV-2 IgM and IgG will be measured from blood samples between 3-6 weeks after the 2nd dose of vaccination

SUMMARY:
This study aimed to investigate the effectiveness of CoronaVac vaccine, which is more than 90% protective in healthy people, in cancer patients receiving active chemotherapy. In this study, to collect information to measure the amount of antibodies produced by the vaccine in the blood of volunteers with the CoronoVac vaccine and to compare it with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Group 1

  1. 18 years old and above
  2. Having completed two doses of CoronoVac vaccine on time
  3. Those with a pathological diagnosis of breast cancer or lung cancer
  4. Being the first dose of vaccine during active chemotherapy period
  5. Ecog performance score 0-1
  6. Patients who signed the informed voluntary consent form
* Group 2

  1. Over 18 years old
  2. Ecog performance score is 0-1
  3. Those who have completed 2 doses of coronovac vaccine within the recommended period
  4. Volunteer who signed the informed consent form

Exclusion Criteria:

* For all groups

  1. Being confirmed or suspected covid-19 before vaccination
  2. Symptomatic covid-19 infection
  3. Being addicted to alcohol or drugs
  4. Having a fever of 37.8 ° C as a suspect before vaccination
  5. Aspleni

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast or lung cancer patients receiving active chemotherapy and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 291 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Antibody levels above the defined cut-off | Between the third and sixth weeks after the second dose of vaccine
  SARS-CoV-2 IgG II ≥ 50.0 AU/ml (positive) and SARSCoV- 2 IgM >1 (positive)

CONTACTS AND LOCATIONS:
Overall Officials: Erdoğan Selçuk Şeber, Asoc.prof, Study Chair — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi İç Hastalıkları ABD, Tıbbi Onkoloji; Halil Taşkaynatan, Asoc.prof, Principal Investigator — İzmir Özel Ege Şehir Hastanesi; Özkan Alan, MD, Principal Investigator — Tekirdağ Dr. İsmail Fehmi Cumalıoğlu Şehir Hastanesi; Üyesi Sonat Pınar Kara, MD, Principal Investigator — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi İç Hastalıkları ABD, İç Hastalıkları; Aliye Çelikkol, MD, Principal Investigator — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi Tıbbi Biyokimya ABD,; Okan Avcı, MD, Principal Investigator — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi İç Hastalıkları ABD, Tıbbi Onkoloji; Eyyüp Çavdar, MD, Principal Investigator — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi İç Hastalıkları ABD, Tıbbi Onkoloji; Kubilay Karaboyun, MD, Principal Investigator — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi İç Hastalıkları ABD, Tıbbi Onkoloji; Berna Erdal, DR, Principal Investigator — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi Mikrobiyoloji ABD; Yakup İriağaç, MD, Study Director — Tekirdağ Namık Kemal Üniversitesi, Tıp Fakültesi İç Hastalıkları ABD, Tıbbi Onkoloji
Locations (1):
- Tekirdağ Namık Kemal ÜNiversitesi, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided